CLINICAL TRIAL: NCT06278311
Title: Association of Presenting Symptoms and Diagnosis, With Urinary Mycotoxins, Metals, Polyfluorinated Alkyl Substance (PFAS) and Environmental Toxins - A Prospective Study in an Urban Gastroenterology Practice
Brief Title: Correlation of Toxins With Gastrointestinal (GI) and Overall Health
Status: Not yet recruiting | Type: Observational
Sponsor: Vibrant America Clinical Lab (Industry)
Collaborators: Los Angeles Integrative Gastroenterology and Nutrition, Inc (Unknown)
Responsible Party: Sponsor
Other Study IDs: 20235761
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Gastrointestinal Diseases
Keywords: Gastrointestinal symptoms; Toxins; Environmental Toxins; Heavy metals; PFAS; Mycotoxins
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: This group will include individuals presenting with digestive and/or non-digestive symptoms or conditions and whose medical evaluation necessitates 'toxin assessment.'
- Healthy controls: This group will include individuals not presenting with digestive and/or non-digestive symptoms or conditions and who volunteer to provide urine samples for 'toxin assessment.'

SUMMARY:
The goal of this observational study is to evaluate the levels of urinary environmental toxins, heavy metals, PFAS and mycotoxins with gastrointestinal (GI) and overall health.

DETAILED DESCRIPTION:
This study aims to use urine samples to understand the effect of toxins such as environmental toxins, heavy metals, PFAS and mycotoxins on GI and overall health. Urine samples will be tested using mass-spectroscopy-based techniques. A 'total toxicity score' will be calculated based on the urine analysis of toxins. A 'symptoms score' will be determined using the 'Symptom History' form which will be used to assess the patient's GI conditions. Additionally, a 'diagnosis score' will be calculated from the diagnosis generated in the electronic medical record (EMR). The determined 'total toxicity score' will be correlated with the 'symptoms score' and the 'diagnosis score.' The observations from this study will help us understand the potential effect of environmental toxins, heavy metals, PFAS and mycotoxins on GI and overall health.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from gastrointestinal and/or other symptoms
* Patients willing to provide urine samples
* Patients willing to provide consent

Exclusion Criteria:

* Use of antibiotics 2 weeks prior to the study
* Patients unwilling to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient group will include individuals presenting with digestive and/or non-digestive symptoms or conditions and whose medical evaluation includes 'toxin assessment,' as determined by the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the Total Toxicity score | 1 year
  Mass spectroscopy-based techniques will be used to test participants' urine samples for environmental toxins, heavy metals, PFAS, and mycotoxins. A 'total toxicity score' will be calculated based on the results obtained from the urine analysis of these toxins. The range for total toxicity score lies between 0 (none) to 232 (severe). Higher scores correspond with worse outcomes.
Determination of the Symptom score | 1 year
  The Symptom History Form is a 90-item questionnaire that will assess participants' digestive and non-digestive symptoms. The scale ranges from 0 (absent) to 1 (present). This form will help determine the 'symptom score.'
Determination of the Diagnosis score | 1 year
  A diagnosis will be selected by the clinician as part of the medical evaluation during the follow-up patient visit. Diagnosis may be "confirmed," "suspected," or "rule out" all as part of a practitioner's clinical impressions. Each diagnosis score will be presented in the form of an International Classification of Diseases (ICD)-10 code. This will help determine the 'diagnosis score,' which applies only to the patient group.

SECONDARY OUTCOMES:
Determination of individual scores | 1 year
  Based on the urine analysis, individual scores for environmental toxins, heavy metals, PFAS, and mycotoxins will be determined. The individual score ranges are as follows: Environmental toxins: 0 (none) to 78 (severe); Heavy metals: 0 (none) to 40 (severe); PFAS: 0 (none) to 52 (severe); Mycotoxins: 0 (none) to 62 (severe). In all cases, higher scores correspond with worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Farshid S Rahbar, MD, Principal Investigator — Los Angeles Integrative Gastroenterology and Nutrition, Inc; Hari K Krishnamurthy, MS, Principal Investigator — Vibrant America Clinical Lab
Locations (2):
- United States (2):
  - Los Angeles Integrative Gastroenterology and Nutrition, Inc, Los Angeles, California
  - Vibrant America Clinical Lab, Santa Clara, California

IPD SHARING:
Plan to Share IPD: No